CLINICAL TRIAL: NCT01716507
Title: A Prospective, Randomized Study Comparing 23-gauge and 20-gauge Pars Plana Vitrectomy for Repair of Pseudophakic Rhegmatogenous Retinal Detachments
Brief Title: 23 Gauge and 20 Gauge Vitrectomy for Rhegmatogenous Retinal Detachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23VS20RD; IRB08858 (Other: WillsEyeIRB)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Retinal Detachment
Keywords: RRD; Rhegmatogenous; Retinal; Detachment; PPV; Pars Plana Vitrectomy; Gauge
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 gauge pars plana vitrectomy (Other): 20 gauge pars plana vitrectomy for retinal detachment repair
  Interventions: Procedure: Retinal Detachment repair
- 23 gauge pars plana vitrectomy (Other): 23 gauge pars plana vitrectomy for retinal detachment repair
  Interventions: Procedure: Retinal Detachment repair

INTERVENTIONS:
Procedure: Retinal Detachment repair — Comparing 23 gauge vs 20 gauge pars plana vitrectomy.

SUMMARY:
This study is a comparison (23 gauge vs 20 gauge instrumentation) of surgical instrumentation for retinal detachment repair.

DETAILED DESCRIPTION:
The majority of studies on PPV for PRD up to this time have used 20-gauge instrumentation. Currently, both 23-gauge and 20-gauge instrumentation are commercially available for PPV. No studies have reported the efficacy of 23-gauge PPV compared to 20-gauge PPV for primary pseudophakic RRD. As a result, many retinal surgeons choose the modality based on personal preference.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent and comply with study assessments for the full duration of the study.
* Presence of retinal detachment with history of cataract surgery.
* Vision of hand motion or better.

Exclusion Criteria:

* Presence of a very large tear or type of retinal detachment usually a result of trauma.
* Prior eye surgery except for cataract surgery.
* Presence of significant scar tissue.
* Presence of retinal detachment due to hole in the macula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assess the initial retinal reattachment rates by comparing the percentages/amount. | 1 Year

SECONDARY OUTCOMES:
Change in best-corrected visual acuity by comparing letters read. | 6 months
  To determine the change in best-corrected visual acuity (BCVA) at the pre-operative visit compared to the 6 month post-operative visit
Reattachment rates with 23 gauge and 20 gauge PPV by comparing the amount. | 1 year
  To determine the final retinal reattachment rates with 23-gauge and 20-gauge PPV if multiple surgeries are required.
Operating time for 23 gauge versus 20 gauge PPV (time measurement) | 1 day- Day of surgery
  This will be done to determine operating times for 23-gauge versus 20-gauge PPV for primary repair of PRD.

OTHER OUTCOMES:
Compare rates of intraoperative and postoperative complications by comparing the amount and severity of these complications. | 1 year
  To describe and compare rates of intraoperative and postoperative complications with 23-gauge versus 20-gauge PPV for primary repair of PRD, including but not limited to post-operative hypotony, choroidal detachment, proliferative vitreoretinopathy, and endophthalmitis.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye
Locations (1):
- Mid Atlantic Retina, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No